CLINICAL TRIAL: NCT02027389
Title: Clinical and Economic Impact of a Rapid Test for Detection of Methicillin-resistant Staphylococcus Aureus (MRSA) From Sterile Sites (the Alere™ PBP2a)
Brief Title: Impact of Rapid Detection of MRSA
Status: Withdrawn | Type: Observational
Why Stopped: personnel change, unable to continue study
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ritu Banerjee, M.D., Ph.D., Associate Professor, Mayo Clinic
Other Study IDs: 13-008045
Record Dates: First submitted 2013-12-27; First posted 2014-01-06 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Staphylococcus Aureus Infections
Keywords: MSSA, MRSA
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control: Patients with growth of S. aureus from sterile site cultures between Sept 15, 2012 - Dec 31, 2012. No rapid testing was performed, and standard bacterial culture and susceptibility testing was done.
- intervention: Patients with growth of S. aureus from sterile site cultures between Sept 15, 2013 - Dec 31, 2013. Rapid PBP2a testing was performed along with pharmacist notification of service if modification to therapy needed based on rapid test results.

SUMMARY:
The objective of this study is to evaluate the impact of the Alere™ PBP2a test combined with pharmacist review of antimicrobial therapy, on clinical outcomes and cost in hospitalized patients with sterile site S. aureus infection.

ELIGIBILITY:
Inclusion criteria:

1. Inpatients (adults and children) at Mayo Clinic, Rochester with sterile source S. aureus cultures (both control and intervention periods)
2. Above, with rapid PBP2a testing (intervention period only).

Exclusion criteria:

1. Patients with polymicrobial cultures (i.e., growth of S. aureus plus other organisms in the culture).
2. Patients who have not provided MN authorization to use their medical records for research.
3. Patients who have had the FilmArray Blood culture identification diagnostic test performed on an index S. aureus blood culture.
4. Patients who have had a sterile source S. aureus culture within the prior 30 days.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients (adults and children) at Mayo Clinic, Rochester with sterile source S. aureus cultures between Sept 15, 2012 - Dec 31, 2012 (control) and Sept 15, 2013 - Dec 31, 2013 (intervention)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Time (hours) to optimal antimicrobial therapy for patients with MSSA and MRSA infections in the pre-intervention and post-intervention periods | within first 7 days of culture result

SECONDARY OUTCOMES:
Time (in hours) to identification of MRSA. | within first 3 days of culture result
Vancomycin days of therapy following S. aureus culture result | during the 2 weeks following culture result

OTHER OUTCOMES:
Proportion of patients with MSSA infection who are switched from an MRSA-active drug to an MSSA-active drug . | within 48 hours of Gram-stain result
Duration of bacteremia in patients with MSSA or MRSA bloodstream infections | within first 30 days of culture result
Time to contact isolation in patients with MRSA infections | within first 7 days of culture result
Length of hospitalization | from time of culture result to hospital discharge, an expected average duration of 4 weeks
Total healthcare costs (broken down by bed, laboratory, and pharmacy costs). | from time of culture result to time of hospital discharge, an expected average duration of 4 weeks
  participants will be followed for the duration of hospital stay following positive culture result, an expected average of 4 weeks.
Proportion of patients where a electronic (P-care) rule flagged for discordant therapy for the PBP2a result | within first 3 days after culture result
Proportion of patients where the pharmacist contacted the service to modify therapy | wihtin first 7 days after culture result

CONTACTS AND LOCATIONS:
Overall Officials: Ritu Banerjee, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States